CLINICAL TRIAL: NCT04359121
Title: COVID-19 and the Developement of Phobic Fears of Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 32-354 ex 19/20
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Physicians: Questionnaires
  Interventions: Other: Questionnaires for specific phobia
- Medical staff: Questionnaires
  Interventions: Other: Questionnaires for specific phobia
- General public: Questionnaires
  Interventions: Other: Questionnaires for specific phobia
- Patients with psychiatric disorders: Questionnaires
  Interventions: Other: Questionnaires for specific phobia

INTERVENTIONS:
Other: Questionnaires for specific phobia — Questionnaires will be used.

SUMMARY:
A lot of people suffer from phobias. Phobias concerning certain diseases are not rare. This study will examine whether the COVID-19 (Coronavirus Disease) crisis was able to rise phobias in people and if those with preexisting phobias or fears were more likely to develop a phobia concerning COVID. It will look at different subtypes - physicians, medical staff, general public (not medically affiliated) and patients with psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Person gives written consent
* Persons between 18-90 years of age (men and women)
* No positive COVID infection known at time of first examination

Exclusion Criteria:

* Dementia, Delirium (not able to give consent)
* Not fulfilling the inclusion criteria
* COVID infection known at first examination point

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: physicians, medical staff, general public, patients with psychiatric disorders
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Development of phobias | 2 years
  Specific Phobia Questionnaire (SPQ): The SPQ consists of 43 items, each rated using a 5-point Likert scale on two dimensions: (1) level of fear, with scores ranging from 0 (no fear) to 4 (extreme fear) and (2) extent to which the fear interferes with one's daily life, with scores ranging from 0 (no interference) to 4 (extreme interference). The SPQ is scored by combining fear ratings of each Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) specific phobia type.
  Severity Measure for Specific Phobia-Adult: The total score can range from 0 to 40 with higher scores indicating greater severity of specific phobia.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baranyi, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No